CLINICAL TRIAL: NCT04713033
Title: Computational Cranial and Cervical Muscle Network in Normal and Disordered Voice
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-01770
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Dysphonia
MeSH Terms: conditions — Dysphonia | interventions — Electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vocally Healthy Controls: Patients will undergo a single experiment to quantify cervical-cranial muscle network patterns during vocal tasks at baseline and after a vocally fatiguing vocal loading task (loud reading) and typical swallowing task.
  Interventions: Diagnostic Test: surface electromyogram (sEMG); Diagnostic Test: flexible laryngoscopy
- Muscle Tension Dysphonia Patients: Patients with muscle tension dysphonia will be measured at baseline and approximately 2 months after their baseline visit following a standard course of voice therapy.
  Interventions: Diagnostic Test: surface electromyogram (sEMG)
- Unilateral Vocal Fold Paralysis Patients: Patients with unilateral vocal fold paralysis will be measured at baseline approximately 2 weeks after receiving a vocal fold medialization injection.
  Interventions: Diagnostic Test: surface electromyogram (sEMG)

INTERVENTIONS:
Diagnostic Test: surface electromyogram (sEMG) — A device that measures electrical signals from your skin will be connected to those stickers and will make a graph that is characteristic to your vocal function.
  Other Names: Trigno Wireless Biofeedback System
Diagnostic Test: flexible laryngoscopy — A device that examines the throat and nasal passages. The flexible laryngoscope or "scope" consists of an eyepiece and a fiber-optic light enclosed in a thin, flexible tube. The scope looks like a strand of black spaghetti with a tiny light on the end of it. The scope is inserted through the nose, and can be moved around to help the doctor see all areas of the nasal passages and throat.
  Other Names: PENTAX Medical ENT Video Imaging System
  Groups: Vocally Healthy Controls

SUMMARY:
The long-term goal is to transform the diagnosis and treatment of dysphonia by elucidating cervical and cranial neuromuscular mechanisms underlying typical and disordered voicing. The overall objective of this application is to propose and evaluate a novel objective spectrotemporal diagnostic tool measuring functional cervical-cranial muscle network activity in typical and disordered speakers.The purpose of this study is to improve our understanding of how the vocal tract and the muscles of the larynx and the head work at baseline and after vocal fatigue.

DETAILED DESCRIPTION:
Three experiments will be conducted over the 2-year award period. Experiment 1 (Aim 1) will utilize a 16-channel EMG array to characterize cervical-cranial muscle activity networks in typical speakers at baseline and after a vocal loading task. Aim 2 will quantify how cervical muscle networks are perturbed in patients with two different types of dysphonia and examine if standard-of-care treatment restores cervical-cranial muscle networks to more typical states. In Experiment 2 (Aim 2), we will measure muscle networks in patients with muscle tension dysphonia before and after a course of voice therapy. Patients with muscle tension dysphonia represent an intact butpotentially maladaptive network. In Experiment 3 (Aim 2), we will measure patients with unilateral vocal fold paralysis, representing a neurologically impaired network, before and after a vocal fold injection medialization procedure.

ELIGIBILITY:
Inclusion Criteria:

Experimental Group

* Age >18 years;
* Patient cohorts diagnosed with muscle tension dysphonia with a recommended treatment of voice therapy.
* Patient cohorts diagnosed with unilateral vocal cord paralysis with a recommended treatment of vocal fold injection medialization.
* Willingness to complete all clinical/research assessments
* Ability to give informed consent

(Control Group)

* Age >18 years;
* Absence of any organic vocal lesion as determined on flexible laryngoscopy.
* Willingness to complete all clinical/research assessments
* Ability to give informed consent

Exclusion Criteria:

Experimental Group:

* Any contraindication for wearing the device, such as a known or reported (at any time including during the study):
* allergy;
* history of head and neck surgery in the past 3 months;
* presence of open wound or/and ulcer in close proximity to sEMG sensors;
* 'smart' implant with a microcontroller (such as a pain pump or nerve stimulator);
* participation in additional clinical research studies using investigational treatments.

Control group:

* Any contraindication for wearing the device, such as a known or reported (at any time including during the study) allergy;
* Abnormal laryngeal structure and function as determined via laryngeal endoscopic exam;
* History of head and neck surgery in the past 3 months;
* Presence of open wound or/and ulcer in close proximity to sEMG sensors;
* 'Smart' implant with a microcontroller (such as a pain pump or nerve stimulator);
* Participation in additional clinical research studies using investigational treatments.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There will be four cohorts of subjects in the study:
  * Cohort one will comprise vocally healthy controls
  * Cohort two will comprise patients with Muscle Tension Dysphonia
  * Cohort three will comprise patients with unilateral vocal fold paralysis
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Change in Pitch and Loudness levels in vocal tasks | Baseline visit, 2 week visit, 2 months visit
  Both at baseline and after a vocal loading task, muscle network activity using sEMG will be measured in a variety of vocal tasks outlined above in Table 1 to explore the muscle network across different vocal demands and pitch and loudness levels. The pitch and loudness of each task produced at baseline by each participant will be calculated, and visual feedback will be provided to participants using the Real-Time Pitch module of the Computerized Speech Lab (Pentax, Montvale, NJ) to help them reproduce similar pitch and loudness levels during post-loading recordings.
Change in Vocal loading task | Baseline visit, 2 week visit, 2 months visit
  After baseline sEMG measurements, vocal fatigue will be induced using a vocal loading task of reading in the presence of 70-dB background noise, as described in Sundarrajan 51 The duration of reading that induces self-perceived vocal fatigue varies among vocally-healthy individuals.52 Therefore, we will use the CR10 Physical Exertion Scale adapted for vocal effort to have participants rate their self-perceived participant reported
Change in Phonatory Effort (PPE) | Baseline visit, 2 week visit, 2 months visit
  Phonatory Effort (PPE) while reading the first section of "The Rainbow Passage" at up to four time points during the load task. The vocal loading task will end after participants report an increase of at least 2 points in PPE.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Johnson, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data Upon reasonable request. Requests should be directed to achlae01@nyu.edu. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT04713033/ICF_000.pdf